CLINICAL TRIAL: NCT05539937
Title: Prospective Evaluation of the Quality of Life of Elderly Patients Undergoing Transfemoral Percutanous Aortic Valve Replacement (TAVI) for the Treatment of Severe Aortic Stenosis. (TAVI QdV)
Brief Title: Prospective Evaluation of the Quality of Life of Elderly Patients Undergoing Transfemoral Percutanous Aortic Valve Replacement (TAVI) for the Treatment of Severe Aortic Stenosis.
Acronym: TAVI QdV
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Collaborators: Belledonne clinic (Unknown); European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00820-43
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Quality of Life; Aortic Valve Replacement; Transfemoral Approach

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with percutaneous aortic valve replacement via the transfemoral approach
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire — Before TAVI, 30 days, 6 months and twelve months after TAVI, patients will answer TASQ questionnaire,

SUMMARY:
In order to overcome the shortcomings of the assessment questionnaires currently available on the assessment of overall quality of life, the "Toronto Aortic Stenosis Quality of Life Questionnaire" (TASQ) was developed as a specific assessment tool for the impact of severe aortic stenosis in elderly patients, through 16 questions covering 5 domains: symptoms and physical limitations, emotional impact and expectations following TAVI, as well as social limitations incurred.

A better knowledge and understanding of the clinical outcomes and quality of life of elderly patients with severe symptomatic aortic stenosis at 12 months of follow-up of a TAVI procedure would further optimize the clinical decision-making process and patient selection who will benefit the most from this intervention in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, over 18 years old,
* All patients who will have transfemoral percutaneous aortic valve replacement (TAVI) with implantation of a valve delivered on a balloon,
* Patient able to understand the study, and answer the TASQ questionnaire,
* Affiliation to a social security scheme or beneficiary of such a scheme,
* Patient having signed the free and informed consent.

Exclusion Criteria:

* Minor,
* Disorder of comprehension and/or expression,
* Patients unable to answer questions due to an underlying cognitive deficit or physical disability,
* Patients treated with a self-expanding valve,
* Refusal to participate in the study,
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision,
* Pregnant, parturient, or breast-feeding patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who will have benefited of a transfemoral percutaneous aortic valve replacement; male or femal over 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in the TASQ global score 12 months after TAVI compared to the TASQ global score before TAVI | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jean-François Oudet, La Rochette, France